CLINICAL TRIAL: NCT01040819
Title: Does Pioglitazone Increase the Production of Prostacyclin (PGI2) and/or 15-EPI-Lipoxin A4 in Humans With Diabetes Mellitus Type 2?
Brief Title: Does Pioglitazone Increase the Production of 15-EPI-Lipoxin A4?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Yochai Birnbaum, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24253
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; 6-Ketoprostaglandin F1 alpha; 15-epi-lipoxin A4; Thiazolidinediones; Pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone 15 mg (Experimental): Patients will receive PIO 15 mg/d for two months. Serum and urine samples for 6-keto-PGF1a and 15-epi-lipoxin A4 will be taken at baseline, one month and 2 months.
  Interventions: Drug: Pioglitazone
- Pioglitazone 30 mg/d (Experimental): Patients will receive PIO 15 mg/d for one month. Then, dose will be increased to 30 mg/d for an additional month. Serum and urine samples for 6-keto-PGF1a and 15-epi-lipoxin A4 will be taken at baseline, one month and 2 months.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Patients will receive PIO 15 mg/d for one month, then 55 patients continue with the same dose for one additional month, and in 55 patients the dose will be increased to 30 mg/d for an additional one month. Other non-diabetes drugs should not be changed. Other hypoglycemic agents, including insulin may be adjusted, if clinically indicated. NSAID, COX2 inhibitors, aspirin >162 mg/d, steroids and prostaglandin analogs will be prohibited.
  Other Names: Actos

SUMMARY:
Type-2 diabetes mellitus is a public health concern. Patients with type 2 diabetes mellitus are at high risk of developing cardiovascular complications. Diabetic patients are two to four-times more likely to develope cardiovascular disease. The mortality of diabetic patients with cardiovascular disease is much higher than in non-diabetic matched patients with cardiovascular disease. Recently, it has become apparent that not all anti-diabetic drugs have the same effect on the progression of atherosclerosis and on cardiovascular outcomes. There is a great need to understand the potential protective mechanisms of the various anti-diabetic drugs in order to decrease their risk for cardiovascular morbidity and mortality. In addition to increasing insulin sensitivity, Pioglitazone (PIO) has anti-inflammatory properties. However, the underlying mechanisms of these anti-inflammatory (and probably anti-atherosclerotic) effects of PIO are unknown. We have shown in the rat that 3-day pretreatment with PIO increases myocardial cyclooxygenase-2 (COX2) activity and levels of both 6-keto-PGF1a, the stable metabolite of prostacyclin (PGI2) and 15-epi-lipoxin A4, a lipid mediator with a strong anti-inflammatory properties. Prostacyclin inhibits platelet aggregation and causes vasodilatation. Increased levels of 6-keto-PGF1a and 15-epi-lipoxin A4 may thus be the explanation for the anti-inflammatory and anti-atherosclerosis effects of PIO. Several clinical studies have shown that COX2 inhibition is associated with increased cardiovascular events. Thus, augmenting COX2 activity and the production of prostacyclin and 15-epi-lipoxin A4 may have potential favorable effects. The purpose of the study is to test whether PIO therapy is associated with an increase in serum and/or urine levels of 6-keto-PGF1a and 15-epi-lipoxin A4 in patients with diabetes mellitus type 2.

DETAILED DESCRIPTION:
Type-2 diabetes mellitus is a public health concern. According to the World health organization (WHO), diabetes mellitus affects more than 180 million people worldwide. Type 2 diabetes mellitus accounts for 80-95% of diabetes cases in developed countries and a higher proportion in developing countries (IDF 2006). Patients with type 2 diabetes mellitus are at high risk of developing cardiovascular complications. Diabetic patients are two to four-times more likely to develope cardiovascular disease. The mortality of diabetic patients with cardiovascular disease is much higher than in non-diabetic matched patients with cardiovascular disease. Recently, it has become apparent that not all anti-diabetic drugs have the same effect on the progression of atherosclerosis and on cardiovascular outcomes. There is a great need to understand the potential protective mechanisms of the various anti-diabetic drugs in order to decrease their risk for cardiovascular morbidity and mortality. In addition to increasing insulin sensitivity, Pioglitazone (PIO) has anti-inflammatory properties. Several studies have suggested that PIO decreases serum markers of inflammation including C-reactive protein (CRP). However, the underlying mechanisms of these anti-inflammatory (and probably anti-atherosclerotic) effects of PIO are unknown. We have shown in the rat that 3-day pretreatment with PIO increases myocardial cyclooxygenase-2 (COX2) activity and levels of both 6-keto-PGF1a, the stable metabolite of prostacyclin (PGI2) and 15-epi-lipoxin A4, a lipid mediator with a strong anti-inflammatory properties. Prostacyclin inhibits platelet aggregation and causes vasodilatation. Increased levels of 6-keto-PGF1a and 15-epi-lipoxin A4 may thus be the explanation for the anti-inflammatory and anti-atherosclerosis effects of PIO. Several clinical studies have shown that COX2 inhibition is associated with increased cardiovascular events. Thus, augmenting COX2 activity and the production of prostacyclin and 15-epi-lipoxin A4 may have potential favorable effects. The purpose of the study is to test whether PIO therapy is associated with an increase in serum and/or urine levels of 6-keto-PGF1a and 15-epi-lipoxin A4 in patients with diabetes mellitus type 2.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women > 21 years old with type 2 diabetes Mellitus and otherwise stable medical conditions

Exclusion Criteria:

1. Serum creatinine >= 1.5 mg/dl and/or renal failure
2. NYHA class III or IV heart failure
3. Known intolerance to TZD
4. Current use of NSAID, COX-2 inhibitors, steroids (oral, topical and inhalation) or immunosuppressive therapy
5. Aspirin > 162 mg/d
6. Recent myocardial infarction, ACS, or stroke <=3 months)
7. Significant comorbid conditions such as: cancer (not cured), end stage renal disease, severe obstructive lung disease, cirrhosis, etc)
8. Recent (<1 month) infection
9. Recent CABG or PCI (<3 months)
10. Use of prostaglandin analogs (i.e., iloprost)
11. Active inflammatory disease
12. Current use of TZD
13. Pregnancy
14. Osteoporosis or high risk for bone fracture. Use of other antihyperglycemic agents is not an exclusion criterion. HbA1c and glucose levels will not restrict enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yochai Birnbaum, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor Clinics, Houston, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye Y, Lin Y, Perez-Polo JR, Uretsky BF, Ye Z, Tieu BC, Birnbaum Y. Phosphorylation of 5-lipoxygenase at ser523 by protein kinase A determines whether pioglitazone and atorvastatin induce proinflammatory leukotriene B4 or anti-inflammatory 15-epi-lipoxin a4 production. J Immunol. 2008 Sep 1;181(5):3515-23. doi: 10.4049/jimmunol.181.5.3515. PMID 18714024
- [Background] Birnbaum Y, Ye Y, Lin Y, Freeberg SY, Huang MH, Perez-Polo JR, Uretsky BF. Aspirin augments 15-epi-lipoxin A4 production by lipopolysaccharide, but blocks the pioglitazone and atorvastatin induction of 15-epi-lipoxin A4 in the rat heart. Prostaglandins Other Lipid Mediat. 2007 Feb;83(1-2):89-98. doi: 10.1016/j.prostaglandins.2006.10.003. Epub 2006 Nov 7. PMID 17259075
- [Background] Birnbaum Y, Ye Y, Lin Y, Freeberg SY, Nishi SP, Martinez JD, Huang MH, Uretsky BF, Perez-Polo JR. Augmentation of myocardial production of 15-epi-lipoxin-a4 by pioglitazone and atorvastatin in the rat. Circulation. 2006 Aug 29;114(9):929-35. doi: 10.1161/CIRCULATIONAHA.106.629907. Epub 2006 Aug 14. PMID 16908763

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone 15 mg: Patients will receive PIO 15 mg/d for two months. Serum and urine samples for 6-keto-PGF1a and 15-epi-lipoxin A4 will be taken at baseline, one month and 2 months.
  Pioglitazone: Patients will receive PIO 15 mg/d for one month, then 55 patients will continue with the same dose for one additional month, and in 55 patients the dose will be increased to 30 mg/d for an additional one month. While on PIO, other non-diabetes drugs should not be changed, unless emergency. Other hypoglycemic agents, including insulin may be adjusted, if clinically indicated. NSAID, COX2 inhibitors, aspirin >162 mg/d, steroids and prostaglandin analogs will be prohibited. At baseline, and after 1, and 2 months of treatment the following samples will be taken: 1. Serum for lipid profile, ALT, AST, CK, creatinine, BUN, glucose, HbA1c (the biochemistry laboratory at UTMB) 2. Serum for 6-keto-PGF1a and 15-epi-lipoxin A4 3. Serum for hs-CRP 4. Urine for creatinine, 6-keto-PGF1a and 15-epi-lipoxin A4
Period: Overall Study
Arm/Group | Pioglitazone 15 mg | Pioglitazone 30 mg/d
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone 15 mg | Pioglitazone 30 mg/d | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (4) | 58 (6) | 56 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Plasma 15-epi-lipoxin A4
Description: Plasma 15-epi-LXA4 levels
Time Frame: 2 months
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Pioglitazone 15 mg | Pioglitazone 30 mg/d
Number analyzed (Participants) | 13 | 12
ng/ml | 1.05 (0.08) | 1.08 (0.12)

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Pioglitazone 15 mg | Pioglitazone 30 mg/d
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No